CLINICAL TRIAL: NCT02858245
Title: A Feasibility Registry on Use of Actigraphy Monitoring in Degenerative Mitral Regurgitation (DMR) Subjects Receiving the MitraClip® Device
Brief Title: A Feasibility Registry of Actigraphy Monitoring in Degenerative Mitral Regurgitation Subjects Receiving the MitraClip® Device
Acronym: VELOCITY
Status: Terminated | Type: Observational
Why Stopped: Study has been terminated due to small sample size
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-6001
Record Dates: First submitted 2016-07-20; First posted 2016-08-08 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2017-05

CONDITIONS: Mitral Regurgitation
Keywords: MitraClip; Structural Heart Failure; Degenerative Mitral Regurgitation (DMR); Actigraphy
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Commercial MitraClip® patients: Patients with Degenerative Mitral Regurgitation receiving MitraClip® Device
  Interventions: Other: No intervention - registry

INTERVENTIONS:
Other: No intervention - registry

SUMMARY:
A prospective, open-label, and multi-centered feasibility registry.

DETAILED DESCRIPTION:
This is a prospective, open-label, and multi-centered feasibility registry (single arm study). Approximately 36 subjects with prohibitive risk degenerative mitral regurgitation (DMR) who receive at least 1 commercial MitraClip will be registered at up to 10 US sites.

ELIGIBILITY:
Inclusion Criteria:

* Subject must consent to receiving the MitraClip device
* Subject must consent, be able, and commit to wearing the Actiwatch continuously for approximately 7 months
* Subject must consent to use of their data from this registry for purposes of exploratory research and publication and presentation

Exclusion Criteria:

* Subject is not a member of vulnerable population
* Subject must not have any disabilities that preclude reliable data collection from the Actiwatch, e.g., epilepsy with uncontrolled recurring episodes, serious stage degenerative/disabling disease (e.g. Parkinson's disease), inability to walk or will require walking aids, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prohibitive risk degenerative mitral regurgitation (DMR) patients who receive at least 1 commercial MitraClip
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Observational change in daily reported activity levels (counts/min) as assessed by actigraphy, from baseline to 30 days post MitraClip implantation | At 30 days
  Phillips Actiwatch Spectrum PRO is the device being used to capture the primary outcome measure

SECONDARY OUTCOMES:
Levels of daily and weekly activity as assessed by actigraphy | Pre-procedure (on day 0)
Levels of daily and weekly activity as assessed by actigraphy | Post-procedure (≤ 7 days)
Levels of daily and weekly activity as assessed by actigraphy | At 30 days
Levels of daily and weekly activity as assessed by actigraphy | At 2 months
Levels of daily and weekly activity as assessed by actigraphy | At 3 months
Levels of daily and weekly activity as assessed by actigraphy | At 4 months
Levels of daily and weekly activity as assessed by actigraphy | At 5 months
Patterns of daily Sleep/Wake by actigraphy | At 6 months
NYHA Functional Class | At Baseline
NYHA Functional Class | At 30 days
Mitral Regurgitation severity | At Baseline
Mitral Regurgitation severity | Post-procedure (≤ 7 days)
Mitral Regurgitation severity | At 30 days
Echocardiographic assessment | At Baseline
Echocardiographic assessment | Post-procedure (≤ 7 days)
Echocardiographic assessment | At 30 days
Distance walked 6 minute walk test (6MWT) | At Baseline
Distance walked 6 minute walk test (6MWT) | At 30 days
Health-related quality of life (QoL) | At Baseline
Health-related quality of life (QoL) | At 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Staehr, MD, Study Director — Abbott Medical Devices
Locations (8):
- United States (8):
  - Banner University Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Baptist Hospital of Miami, Miami, Florida
  - Mayo Foundation for Medical Education and Research, Rochester, Minnesota
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Bon Secours St Mary's Hospital, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No